CLINICAL TRIAL: NCT02830503
Title: Feeding Tube Practices and Colonization of the Preterm Stomach in the First Week of Life: A Randomized Controlled Trial
Brief Title: Feeding Tube Practices and Colonization of the Preterm Stomach in the First Week of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gorm Greisen (Other)
Collaborators: Statens Serum Institut (Other)
Responsible Party: Sponsor-Investigator, Gorm Greisen, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-15021673
Record Dates: First submitted 2016-05-10; First posted 2016-07-13 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Feeding tube daily replacement
  Interventions: Procedure: Feeding tube daily replacement
- Control (No Intervention): Feeding tubes replaced as normal practice in the department (normally once a week).

INTERVENTIONS:
Procedure: Feeding tube daily replacement — Feeding tubes replaced once a day in the first week of life.
  Arms: Intervention

SUMMARY:
Project summary

Rationale

Many NICU's replace their feeding tubes once a week or more rarely in order to avoid disturbing the infants. The researchers discovered that there are high concentrations of potentially pathogenic bacteria in the yield of resident nasogastric feeding tubes, even within one day of use (own data, manuscript submitted). Preterm infants are vulnerable to the colonization of the gut, and development of dysbiosis might lead to necrotizing enterocolitis. The researchers speculate if replacing the resident feeding tube every day and thereby decreasing the amount of potentially pathogenic bacteria given to the infants via the feeding tube will lead to fewer bacteria present in the upper part of the gastrointestinal tract of the infant and hence a reduced competition with probiotic colonization.

Objectives

The investigators plan to conduct an intervention study in premature infants receiving probiotics (< 32 weeks of gestation) where the feeding tube will be replaced every day in the intervention group and once a week (standard practice) in the control group. The main outcome will be bacterial concentration in the stomach after one week of life.

Methods

The study is a prospective, randomized controlled trial in preterm infants. Infants will be randomized to the intervention group in which the tube is replaced every day or the control group which will follow normal practice in the department. The intervention will last one week. The infants will be followed until discharge. The investigators plan to include 11 infants in each group.

Primary outcome

Concentration of bacteria in gastric aspirates on day seven.

ELIGIBILITY:
Inclusion Criteria:

* Under 32 weeks GA at birth
* Admission time considered to be more than seven days
* Signed informed consent within 48 hours after birth

Exclusion Criteria:

* Transfer to another hospital within seven days
* Major gastrointestinal malformations
* No tube feeding within first 48 h of birth

Ages: 1 Hour to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2016-06; Primary Completion 2019-06 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Concentration (CFU/ml) of bacteria in gastric aspirates | on day seven of life

SECONDARY OUTCOMES:
Number of patients with potentially pathogenic bacteria at any concentration in gastric aspirates | day seven of life.
  Qualitative differences between bacteria found in the gastric aspirates of intervention and control group. Potentially pathogenic bacteria= Enterobacteriaceae and S. aureus.
pH (acidity) of gastric aspirates | First week of life
Number of patients with probiotics cultured from gastric aspirates aspirates | First week of life
  Determination of whether probiotic bacteria are detectable in the gastric aspirates, and in which concentration.
Concentration (CFU/ml) of bacteria in maternal milk | First week of life
  Investigate any correlation between maternal milk flora and gastric flora.

CONTACTS AND LOCATIONS:
Overall Officials: Gorm Greisen, Professor, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Neonatology, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Munkstrup C, Krogfelt KA, Greisen G, Juhl SM. Feeding tube practices and the colonisation of the preterm stomach in the first week of life. Dan Med J. 2022 Jul 13;69(8):A06210494. PMID 35959833